CLINICAL TRIAL: NCT00207207
Title: Randomized Trial to Assess the Effect of Using Alternate Site Blood Glucose Testing Versus Finger-Tip Testing on Long-Term Glycemic Control.
Brief Title: Self Monitoring of Blood Glucose With Finger Tip vs. Alternate Site Sampling: Effect on Long Term Glycemic Control
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Caroline Apovian, MD, Boston Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Protocol # 03-004C; Contract #: 233-02-0077
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Diabetes Mellitus
Keywords: Alternate Site; Blood Glucose Testing; Blood Sugar Testing; Hemoglobin A1C
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Alternate site blood glucose testing

SUMMARY:
The objective is to assess the effect of using ASBG (alternate site blood glucose) versus FTBG (finger tip blood glucose) testing on long-term glycemic control in diabetics. Since ASBG measurements appear to lag behind FSBG measurements at times of changing glucose concentration, it is possible that ASBG measurements will yield lower postprandial readings than FTBG, potentially causing a negative impact on long-term control. It is also possible that since ASBG is reportedly more comfortable than FTBG testing, it's use might improve adherence to testing and improve long term control.

DETAILED DESCRIPTION:
Patients undergo an initial screening visit. Inclusion criteria include adults 18 -70 years of age with type II diabetes currently using insulin and recording SMBG measurements. Exclusion criteria include history of severe hypoglycemic episodes, current use of ASBG measurements, serious co-morbid illness or pregnancy. For eligible subjects baseline data including HbA1C is obtained. The goal for enrollment is 176 subjects. Subjects are randomized into either a fingertip or an arm-testing group within strata of baseline HbA1C. Each subject who does not already have one receives a One Touch Ultra® SMBG device. All subjects receive training in the use of this device, but for those in the arm-testing group this includes training on obtaining samples from the forearm. Arm- testing subjects are encouraged to use arm testing as much as possible but to use finger testing if they are not able to obtain a sample from the arm. All subjects are asked to perform SMBG testing before breakfast, before dinner and 2 hours after dinner and to complete diaries of all SMBG readings. At 1, 3 and 5 months after the training visit subjects see a diabetes provider who makes adjustments in the therapeutic regimen based on the SMBG measurements, as they would during routine diabetes management. Diary sheets are then collected and the data they contain is entered into a database. At months 2, 4 and 7 subjects present for a visit to drop off their diary sheets. At months 4 and 7 they have blood drawn for HbA1C measurement. The principal outcome variable is level of diabetic control as measured by 7-month HbA1c. The means for each group will be compared, and we will test the hypothesis that glycemic control as represented by 7-month HbA1C is not worse for the ASBG group than the FTBG group. Secondary outcome variables are compliance with testing and number of hypoglycemic episodes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will include adults 18 -70 years of age with type II diabetes currently using insulin and recording SMBG measurements.

Exclusion Criteria:

Patients will be excluded who have a history of hypoglycemic episodes, within the last two years, requiring urgent medical attention, hypoglycemia resulting in cognitive impairment, a lack of symptoms during hypoglycemic episodes. Subjects will also be excluded who have type I DM as determined by the investigators on a case-by-case basis, subjects who already utilize ASBG measurements or who have serious co-morbid illness (unstable cardiovascular disease, metastatic CA). Pregnant patients will also be excluded because of the more intense diabetic control they require.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174
Dates: Start 2003-07; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Level of diabetic control as measured by 7-month HbA1c.

SECONDARY OUTCOMES:
Compliance with testing.
Number of hypoglycemic episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Apovian, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Ellison JM, Stegmann JM, Colner SL, Michael RH, Sharma MK, Ervin KR, Horwitz DL. Rapid changes in postprandial blood glucose produce concentration differences at finger, forearm, and thigh sampling sites. Diabetes Care. 2002 Jun;25(6):961-4. doi: 10.2337/diacare.25.6.961. PMID 12032099
- [Background] Saaddine JB, Engelgau MM, Beckles GL, Gregg EW, Thompson TJ, Narayan KM. A diabetes report card for the United States: quality of care in the 1990s. Ann Intern Med. 2002 Apr 16;136(8):565-74. doi: 10.7326/0003-4819-136-8-200204160-00005. PMID 11955024
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Fineberg SE, Bergenstal RM, Bernstein RM, Laffel LM, Schwartz SL. Use of an automated device for alternative site blood glucose monitoring. Diabetes Care. 2001 Jul;24(7):1217-20. doi: 10.2337/diacare.24.7.1217. PMID 11423505
- [Background] Kuwa K, Nakayama T, Hoshino T, Tominaga M. Relationships of glucose concentrations in capillary whole blood, venous whole blood and venous plasma. Clin Chim Acta. 2001 May;307(1-2):187-92. doi: 10.1016/s0009-8981(01)00426-0. PMID 11369356
- [Background] Jungheim K, Koschinsky T. Glucose monitoring at the arm: risky delays of hypoglycemia and hyperglycemia detection. Diabetes Care. 2002 Jun;25(6):956-60. doi: 10.2337/diacare.25.6.956. PMID 12032098
- [Background] de Veciana M, Major CA, Morgan MA, Asrat T, Toohey JS, Lien JM, Evans AT. Postprandial versus preprandial blood glucose monitoring in women with gestational diabetes mellitus requiring insulin therapy. N Engl J Med. 1995 Nov 9;333(19):1237-41. doi: 10.1056/NEJM199511093331901. PMID 7565999